CLINICAL TRIAL: NCT04215705
Title: Postoperative Analgesic Efficiency of Quadratus Lumborum Block III Versus Peritubal Local Infiltration in Patients Undergoing exPercutaneous Percutaneous Nephrolithotomy Operation : a Randomized Comparative Study
Brief Title: Quadratus Lumborum Block III Versus Peritubal Local Infiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, simon Halim Armanious, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Post PCNL analgesia
Record Dates: First submitted 2019-12-28; First posted 2020-01-02 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Q (Active Comparator): Patients in this group receive Quadratus Lumborum Block with 20 ml bupivacaine 0.5%
  Interventions: Procedure: Quadratus block versus peritubal local infiltration
- Group L (Active Comparator): Patients in this group receive peritubal local infiltration at 6 and 12 o'clock position with 20ml bupivacaine 0.5%
  Interventions: Procedure: Quadratus block versus peritubal local infiltration

INTERVENTIONS:
Procedure: Quadratus block versus peritubal local infiltration — Quadratus lumborum block III versus peritubal local infiltration in patients undergoing Percutaneous Nephrolithotomy operation

SUMMARY:
Investigators compare post operative analgesic efficacy of peritubal local infiltration versus Quadratus Lumborum Block III . In patients undergoing Percutaneous Nephrolithotomy operation

ELIGIBILITY:
Inclusion Criteria:

* patient with pelvic renal stone less than 2 cm
* Americans society of Anesthesiologists physical status I, II
* BMI<35

Exclusion Criteria:

* patient refusal to participate in the study
* Americans society of Anesthesiologists physical status III or above
* major hepatic, renal or cardiovascular disease
* BMI > 35
* coagulopathy
* psychological disorders.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2020-07-12 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia | 24 hours
  Postoperative pain measured by visual analogue scale from 0 to 10 measured over 24h where 0 is better and 10 means worst pain
Analgesic requirement | 24 hours
  Investigators measured the total dose of morphine consumption in mg over 24hour

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hosptal, Cairo, Abbasya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Upon request from Corresponding Author
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Over 6
  Within 6 month
URL: http://www.synapse.org